CLINICAL TRIAL: NCT00004990
Title: Pulse Dexamethasone in Focal Segmental Glomerulosclerosis
Brief Title: Once-A-Month Steroid Treatment for Patients With Focal Segmental Glomerulosclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000100; 00-DK-0100
Record Dates: First submitted 2000-03-18; First posted 2000-03-20 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-12

CONDITIONS: Glomerulonephritis; Nephrotic Syndrome
Keywords: Nephrotic Syndrome; Steroids; Osteoporosis; Adrenal Suppression; Proteinuria; Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Glomerulonephritis; Nephrotic Syndrome; Osteoporosis; Proteinuria; Glomerulosclerosis, Focal Segmental | interventions — Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone

SUMMARY:
This study will test the safety and effectiveness of a monthly dosing regimen of dexamethasone-a strong steroid medication-to treat patients with focal segmental glomerulosclerosis (FSGS). Patients with this disease have kidney fibrosis (scarring) and proteinuria (excessive excretion of protein in the urine) that, in about half of the patients eventually requires kidney dialysis or transplant. Currently, the most effective treatment for FSGS is high-dose steroids (prednisone) taken daily for 4 to 6 months. However, only about 30 percent of patients respond to this treatment, and it causes serious side effects in many patients. Other drugs, such as cyclosporin and cyclophosphamide, improve proteinuria in even fewer patients (about 10 percent) and also have serious side effects. This study will explore whether a monthly pulse dose of steroids will achieve disease remission with less toxicity.

Adults and children with FSGS who: 1) have not received steroid treatment, or 2) could not tolerate daily steroid treatment, or 3) relapsed after conventional steroid treatment may be eligible for this study. Those enrolled will take dexamethasone by mouth for 4 days every 4 weeks for a total of 8 months. Patients will undergo various tests before treatment starts (baseline), during the course of treatment, and in follow-up visits to evaluate the effects of treatment as follows:

1. Review of kidney biopsy, medical evaluation, measurement of total daily urine protein excretion and kidney function, psychiatric testing for depression or other mood disorder
2. Measurements of blood pressure, blood chemistries and urine protein excretion - monthly during treatment
3. Questionnaire about the effects of treatment, if any, on mood and feelings - monthly during treatment
4. Photographs of the face and body (in underwear or shorts and tank top) to evaluate body fat distribution- baseline and 8 months
5. Eye examinations for cataracts and glaucoma - baseline and 8 months
6. Bone density scan (DEXA scan) of the lower spine and hip - baseline, 4 and 12 months
7. Magnetic resonance imaging (MRI) of the hips
8. Psychological evaluation and quality of life evaluation - baseline, 1, 2 and 8 months
9. Blood tests for adrenal gland function - baseline, 4 and 8 months
10. Blood and urine tests - 10, 12, 15, and 18 months

Patients who achieve remission (whose urine protein levels decrease to normal) before completing the 8 months of dexamethasone will take one more dose and then stop therapy, but continue with follow-up. Patients who achieve remission but relapse may be offered a second course of treatment.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effectiveness and toxicity of an alternative steroid dosing regimen for patients with focal segmental glomerulosclerosis (FSGS), using a pilot study design that will enroll 20 patients. Although the literature reports variable steroid responsiveness, remission rates of up to 30-40 percent have recently been reported in nephrotic adult patients treated with daily prednisone at 1 mg/kg/day for at least 4 months, followed by a taper over 3-4 months. Such a prolonged and aggressive steroid course is fraught with significant morbidity, but this approach has been advocated by some authors because of the poor prognosis for renal survival in nephrotic patients with FSGS who do not achieve remission with steroid treatment. We plan to test an eight month course of high dose steroid therapy administered in monthly pulses instead of daily doses, for comparable efficacy in achieving remission, and for the occurrence of adverse steroid side effects. We plan to enroll patients with nephrotic syndrome due to biopsy-proven FSGS, who have either not been treated, or have responded to conventional steroid dosing regimens and relapsed. We plan to treat them with monthly oral pulses of dexamethasone (40-60 mg/d x 4 days), for 8 months. The primary endpoint will be induction of complete remission, defined as urine protein less than 300 mg/d. Patients will also be evaluated for manifestations of steroid toxicity. Patients will be seen in follow up at intervals up to 24 months following study entry. If this study suggests that remission of nephrotic syndrome can be attained with this regimen, and with an acceptable toxicity profile, we will plan a randomized controlled trial of this regimen compared with daily or alternate day oral steroids.

ELIGIBILITY:
INCLUSION CRITERIA:

Adults and children.

Biopsy proven FSGS, including idiopathic FSGS and collapsing FSGS, but excluding HIV-associated FSGS and secondary FSGS associated with morbid obesity, sickle cell anemia, reflux nephropathy, chronic tubular injury, congenital renal anomalies, and reduced nephron mass.

Glomerular filtration rate will be estimated using 4 variable MDRD GFR equation, which incorporates age, race, gender, and serum creatinine.

If disease has been present less than or equal to 1 year, estimated GFR must be greater than or equal to 40 ml/min.

If disease has been present greater than or equal to 1 year, estimated GFR must be greater than or equal to 60 ml/min.

Nephrotic range proteinuria, defined as urine protein greater than or equal to 3.5 g/1.73 m(2)/d.

Patients who received steroids for FSGS and who entered complete remission but have relapsed with nephrotic range proteinuria will be eligible.

If hypertensive, adequate blood pressure control (target BP less than or equal to 130/80 mm Hg at greater than 75% of measurement in adults).

Patients must have been taking an angiotensin converting enzyme inhibitor or angiotensin receptor antagonist for at least 6 weeks, unless intolerant of these medications.

Women with child-bearing potential must maintain an effective birth control regimen (oral contraceptive, intrauterine device, barrier plus spermicide).

EXCLUSION CRITERIA:

Inability to give informed consent or cooperate with study.

Poorly controlled diabetes (as defined by hemoglobin A1C of greater than or equal to 8.5 on entry screening, or daily insulin requirement of greater than or equal to 100 units) or hypertension (defined as systolic BP consistently greater than 160 and/or diastolic BP consistently greater than 100 on three or more drugs).

Evidence of chronic or occult infection. Specifically, must not have evidence of active hepatitis B, hepatitis C, HIV or untreated mycobacterial infection.

Current or prior use of cytotoxic agents or cyclosporin for FSGS. If previously treated with these agents for a non-renal indication, therapy must have concluded at least 12 months prior to study.

Existence of any other condition which would complicate the implementation or interpretation of the study.

History of steroid-induced psychiatric disorder, known avascular necrosis of hip or symptomatic osteoporosis (e.g., known compression fractures), brittle diabetes mellitus, or glaucoma. Patients with other psychiatric disorders will be evaluated on a case by case basis.

Patients who have been treated with steroids equivalent to 1 mg/kg/day for greater than or equal to 8 weeks without remission will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2000-03; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), Bethesda, Maryland, United States

REFERENCES:
- [Background] Adams DM, Kinney TR, O'Branski-Rupp E, Ware RE. High-dose oral dexamethasone therapy for chronic childhood idiopathic thrombocytopenic purpura. J Pediatr. 1996 Feb;128(2):281-3. doi: 10.1016/s0022-3476(96)70410-9. PMID 8636831
- [Background] Alexanian R, Dimopoulos MA, Delasalle K, Barlogie B. Primary dexamethasone treatment of multiple myeloma. Blood. 1992 Aug 15;80(4):887-90. PMID 1498331
- [Background] Andersen JC. Response of resistant idiopathic thrombocytopenic purpura to pulsed high-dose dexamethasone therapy. N Engl J Med. 1994 Jun 2;330(22):1560-4. doi: 10.1056/NEJM199406023302203. PMID 8177245